CLINICAL TRIAL: NCT06417840
Title: To Evaluate the Impact of Consumption of a Bioactive Compound Extracted From Fermented Yeast on Fasting Blood Glucose Levels in Asian Indians With Pre-diabetes: A Randomized, Double Blinded, Placebo-controlled Parallel Arm Trial
Brief Title: To Evaluate the Impact of Consumption of a Bioactive Compound on Fasting Blood Glucose Levels in Asian Indians With Pre-diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brightseed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1.4/FCDOC/EC/HAO/2024-25
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Control
- N-trans-caffeoyltyramine (NCT) and N-trans-feruloyltyramine (NFT) (Experimental)
  Interventions: Dietary Supplement: N-trans-caffeoyltyramine (NCT) and N-trans-feruloyltyramine (NFT)

INTERVENTIONS:
Dietary Supplement: N-trans-caffeoyltyramine (NCT) and N-trans-feruloyltyramine (NFT) — N-trans-caffeoyltyramine (NCT) and N-trans-feruloyltyramine (NFT) derived via synthetic biology (i.e., fermentation using a recombinant microorganism) to provide a high purity (>85%) form of these compounds that are structurally identical to their naturally occurring counterparts. All ingredients in the encapsulated final test article, including the NCT and NFT, are manufactured under food GMPs and are of suitable quality for use in food, dietary supplements, and specialty nutrition products.
  Arms: N-trans-caffeoyltyramine (NCT) and N-trans-feruloyltyramine (NFT)
Dietary Supplement: Placebo Control — Placebo Control
  Arms: Placebo Control

SUMMARY:
This is randomized placebo controlled, double-blinded, parallel arm study on free living Asian Indians. Eligible subjects will undergo one-week run-in period and subjects will be asked to maintain their usual diet and exercise regime. At the end of the run-in period, subjects fulfilling the inclusion/exclusion criteria at this stage will be randomized either to the intervention arm or control arm using computerized random number tables.

The measured parameters will include, 24-h diet recall, food frequency questionnaire, anthropometry including circumferences, height and weight, and blood parameters including blood glucose (fasting), serum insulin (fasting), HbA1c and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting Blood Glucose between 100-125 mg/dL;
2. and BMI range 25-30 kg/m2;
3. and waist circumference ≥80cm for women and ≥90cm for men;

Exclusion Criteria:

1. Weight loss or gain ≥4.5 kg within 90 days of visit 1.
2. Use of weight loss medications within 90 days of visit 1.
3. History of gastrointestinal surgery (e.g., bariatric surgery) or cosmetic procedures (e.g., liposuction) for weight/fat reducing purposes.
4. Use of dietary supplements or related products that, in the judgment of the Investigator, are likely to markedly affect weight loss or appetite within 30 days of visit 1.
5. History of extreme dietary habits (e.g., Atkins diet, etc.), as judged by the Investigator.
6. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
7. Current medical diagnosis of type 1 or type 2 diabetes mellitus.
8. HbA1c ≥48 mmol/mol (6.5%) as measured at visit 1.
9. History of a chronic gastrointestinal disorder, such as peptic ulcer disease or malabsorption syndrome (mild lactose intolerance or gastroesophageal reflux diseases are acceptable).
10. Signs or symptoms of an active infection of clinical relevance within 5 days of visit 1. The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to visit 1.
11. Is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source document.
12. Any condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.
13. Excessive alcohol consumption (> 2 Drinks, 60 ml of Whisky Per Day).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Glucose | 0, and 28 days
  Blood Glucose Concentration mg/dL

SECONDARY OUTCOMES:
Fasting Blood Insulin | 0, and 28 days
  Blood Insulin Concentration mcIU/mL
HbA1c | 0, and 28 days
  Percent (%) blood HbA1c level
Continuous Glucose Monitoring | 0, and 28 days
  Continuous Blood Glucose Monitoring mg/dL
Total Cholesterol | 0, and 28 days
  Total blood cholesterol mg/dL
Low-density lipoprotein (LDL) cholesterol | 0, and 28 days
  Blood Low-density lipoprotein (LDL) cholesterol mg/dL
High-density lipoprotein (HDL) cholesterol | 0, and 28 days
  Blood High-density lipoprotein (HDL) cholesterol mg/dL
Triglycerides | 0, and 28 days
  Blood Triglycerides mg/dL
Weight | 0, and 28 days
  kg of Body Weight
Height | 0, and 28 days
  Height in meters (m)
Body Mass Index (BMI) | 0, and 28 days
  Body mass index (BMI) measured via weight in kilograms divided by the square of height in meters.
Waist Circumference | 0, and 28 days
  Waist Circumference in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Foundation (India), New Delhi, India